CLINICAL TRIAL: NCT07143422
Title: Sharp Risks in a Time of Crisis: A Study of Needle-Stick Injuries in Eastern Sudan's Healthcare Sector - A Cross-Sectional Study
Brief Title: Sharp Risks in a Time of Crisis: Needle-Stick Injuries in Eastern Sudan Healthcare
Status: Completed | Type: Observational
Sponsor: National Center for Gastroentestinal and Liver Disease (Other)
Responsible Party: Principal Investigator, Ahmed Rafei, Head of Reseach Department, National Center for Gastroentestinal and Liver Disease
Other Study IDs: ncgld
Record Dates: First submitted 2025-08-08; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Needlestick Injuries
Keywords: Needlestick injuries; Health care workers; Safety
MeSH Terms: conditions — Needlestick Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Needle-stick injuries (NSIs) expose healthcare providers to serious bloodborne infections such as HBV, HCV, and HIV. These injuries are prevalent in Africa and worsened by poor training, limited resources, and systemic issues. In Sudan, the ongoing war has intensified healthcare challenges, increasing NSI risks.

Methods: A cross-sectional survey was conducted among doctors and nurses in Eastern Sudan using an interview-based questionnaire. Stratified random sampling ensured proportional representation. Data were analyzed using SPSS (p < 0.05). Ethical approval and informed consent were obtained.

ELIGIBILITY:
Inclusion Criteria:

Doctors who are currently employed and actively working in healthcare facilities such as hospitals and clinics in Kassala and Al Qadarif states, Eastern Sudan.

Nurses who are currently employed and actively working in healthcare facilities such as hospitals and clinics in Kassala and Al Qadarif states, Eastern Sudan.

Healthcare providers who are at risk of needle-stick injuries as part of their routine clinical duties, including procedures involving needles and sharps.

Participants who provide informed consent to take part in the study.

Exclusion Criteria:

Non-clinical staff who do not engage in direct patient care or handling of needles and sharps, such as administrative personnel.

Hygienists and other support staff whose job roles do not involve exposure to needle-stick injuries.

Medical students and trainees who are not fully employed healthcare providers within the facilities at the time of the study.

Individuals who do not consent or refuse to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of doctors and nurses actively employed in healthcare facilities, including hospitals and clinics, within Kassala and Al Qadarif states in Eastern Sudan. These healthcare providers are at risk of needle-stick injuries due to their direct involvement in clinical procedures using needles and sharps. Non-clinical staff, hygienists, medical students, and other personnel not directly involved in patient care or exposure to sharps were excluded. A census with stratified random sampling was used to ensure proportional representation across professions and healthcare settings.
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of Needle-Stick Injuries Among Healthcare Workers | 6 months
  Percentage of healthcare workers reporting ≥1 needle-stick injury.

SECONDARY OUTCOMES:
Proportion of healthcare workers reporting needle-stick injury reporting behavior | 6 months
  Percentage of participants who reported their needle-stick injuries to hospital authorities or occupational health services, assessed by questionnaire.

OTHER OUTCOMES:
Frequency of Needle-Stick Injuries per Participant | 6 months
  Number of needle-stick injuries reported by each participant, categorized as 0, 1-2, or ≥3 incidents.